CLINICAL TRIAL: NCT02880293
Title: Partially HLA-Mismatched Related Donor Hematopoietic Stem Cell Transplantation Using Killer Immunoglobulin Receptor and Human Leukocyte Antigen Based Donor Selection
Brief Title: Haploidentical (Half-matched) Related Donor Stem Cell Transplantation Using Killer Immunoglobulin-like Receptors in Addition to Normal Selection Factors to Determine the Best Donor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-1237
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2023-11

CONDITIONS: Hematologic Malignancy
Keywords: transplant conditioning; KIR/HLA based haploidentical donor selection; allogeneic hematopoietic cell transplantation
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Melphalan; fludarabine; fludarabine phosphate; Thiotepa; Cyclophosphamide; Mesna; Mycophenolic Acid; Filgrastim; Tacrolimus

ARMS (1):
- Patients will undergo donor/recipient bone marrow (Experimental): All patients will undergo haploidentical, allogeneic hematopoietic cell transplantation. Conditioning will consist of fludarabine, melphalan, and thiotepa. Graft versus host disease prophylaxis will be with post-transplant cyclophosphamide in addition to standard tacrolimus and mycophenolate mofetil. Donors will undergo HLA and KIR geno- and allotyping to determine the best donor.
  Interventions: Drug: melphalan; Drug: fludarabine; Drug: thiotepa; Drug: Cyclophosphamide; Drug: Mesna; Drug: Mycophenolate Mofetil; Drug: Filgrastim; Drug: Tacrolimus

INTERVENTIONS:
Drug: melphalan — melphalan (140 mg/m2 IV on day -7)
  Other Names: Alkeran®
Drug: fludarabine — fludarabine (40 mg/m2/d on days -5 through -2)
  Other Names: FLUDARA®
Drug: thiotepa — thiotepa (5 mg/kg IV on day -67)
Drug: Cyclophosphamide — cyclophosphamide (50 mg/kg IV on day +3 and +4)
  Other Names: Cytoxan®
Drug: Mesna
  Other Names: Mesnex®
Drug: Mycophenolate Mofetil — (15 mg/kg PO/IV TID)
  Other Names: CellCept®
Drug: Filgrastim
  Other Names: Neupogen®
Drug: Tacrolimus
  Other Names: Prograf®

SUMMARY:
This study will test whether half matched donors with favorable KIR genes will reduce the risk of cancer recurring after transplant.

ELIGIBILITY:
Inclusion Criteria:

Patients with any of the following hematologic malignancies who are considered to be eligible for allogeneic transplantation:

* Acute lymphoid leukemia (ALL) in first complete remission (CR1) with high riskfor relapse including:
* t(9;22) or detected BCR-ABL1 translocation by genomic methodologies
* BCR-ABL1-Like B-ALL [54] including mutations of IKZF1 or CRLF2
* Translocations or mutations involving 11q23 (MLL) gene.
* Hypodiploid karyotype
* Deletion of 9p
* Loss of 17p or TP53 mutation
* T-lymphocyte lineage antigen expression (T-ALL)
* CNS or other extramedullary involvement
* WBC count >/= 100,000 cells/μL at diagnosis
* Relapsed ALL, biphenotypic/bilineal leukemia, or AML with </= 10% blasts in the bone marrow prior to transplantation
* Acute biphenotypic or bilineal leukemia in first or greater complete remission.
* Acute myeloid leukemia (AML) in CR1 with intermediate or high risk features including:
* Cytogeneic abnormalities associated with myelodysplatic syndrome including abnormalities of chromosome 5 or 7
* History of anti-neoplastic therapy (radiation or chemotherapy)
* Extramedullary involvement
* WBC count >/= 100,00 cells/ul at diagnosis
* Rearrangements or mutations of 11q23 (MLL)
* Abnormalities of chromosome 3
* TP53 mutation or loss of 17p
* Complex or monosomal karyotype
* Normal karyotype with mutations of FLT3, RUNX1, or ASXL1
* Myleodysplastic syndrome, myeloproliferative neoplasms, or MDS/MPN overlap syndrome with:
* International prognostic scoring system risk score of INT-2 or high risk at the time of transplant evaluation
* Any risk category if life-threatening cytopenia exists
* Karyotype or genomic changes that indicate high risk for progression to acute myelogenous leukemia, including abnormalities of chromosome 7 or 3, mutations of TP53, or complex or monosomal karyotype
* Myelofibrosis with DIPSS scores of INT-2 or high risk or any risk category if life threatening cytopenias are present
* Chronic myelomonocytic leukemia (CMML)
* Chronic myeloid leukemia (CML) who have failed or are intolerant to BCR-ABL tyrosine kinase inhibitors
* CML with BCR-ABL mutation consistent with poor response to tyrosine kinase inhibition (e.g. T351 l mutation)
* CML with accelerated or blast phase with <20% blasts after therapy
* Hodgkin lymphoma:
* Relapsed disease with progression after autologous bone marrow transplant or are ineligible for this procedure
* Responding to therapy prior to enrollment
* Non-Hodgkin lymphoma:
* Responding to therapy prior to enrollment
* Progression after autologous bone marrow transplant or are ineligible for this procedure
* Chronic lymphocytic leukemia with high risk disease as defined by the EBMT consensus criteria

  * Patients aged 18 through 69 years old are eligible
  * Patients aged 70-75 with HCT-CI of 0-1 are eligible
  * High risk hematologic malignancies
  * Patients must have Karnofsky performance status >/= 70%
  * Cardiac left ventricular ejection fraction >/= 50% at rest
  * Total bilirubin </= 2 mg/dL, except for patients with Gilbert's syndrome
  * AST and ALT </= 5x ULN unless thought to be disease related
  * Estimated or measured creatinine clearance > 50 mL/min
  * Hemoglobin adjusted pulmonary DLCO >/= 50% of predicted, if Hgb is within normal range, unadjusted DLCO must be >/= 50%

Exclusion Criteria:

* Persons with a HLA matched sibling donor.
* Female patients who are pregnant or breast-feeding
* Persons with an infection that is not responding to antimicrobial therapy
* Persons who are seropositive for HIV.
* Persons with uncontrolled central nervous system malignancy •Persons who do not meet the age and organ function criteria specified above Presence of psychiatric or neurologic disease, or lack of social support that limits the patient's ability to comply with the treatment protocol including supportive care, follow-up, and research tests.
* Prior diagnosis of non-hematologic malignancy within 5 years of planned protocol therapy EXCEPT:

  * Diagnosis of breast ductal carcinoma in situ treated with curative intent
  * Diagnosis of prostate adenocarcinoma with Gleasons score </= 6 treated with curative intent
  * Non-melanomatous skin cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-08-23; Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Shaffer, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Will Undergo Donor/Recipient Bone Marrow: All patients will undergo haploidentical, allogeneic hematopoietic cell transplantation. Conditioning will consist of fludarabine, melphalan, and thiotepa. Graft versus host disease prophylaxis will be with post-transplant cyclophosphamide in addition to standard tacrolimus and mycophenolate mofetil. Donors will undergo HLA and KIR geno- and allotyping to determine the best donor.
  melphalan: melphalan (140 mg/m2 IV on day -7)
  fludarabine: fludarabine (40 mg/m2/d on days -5 through -2)
  thiotepa: thiotepa (5 mg/kg IV on day -67)
  Cyclophosphamide: cyclophosphamide (50 mg/kg IV on day +3 and +4)
  Mesna
  Mycophenolate Mofetil: (15 mg/kg PO/IV TID)
  Filgrastim
  Tacrolimus
Period: Overall Study
Arm/Group | Patients Will Undergo Donor/Recipient Bone Marrow
Started | 44
Completed | 39
Not Completed | 5
Not completed — Inevaluable | 5

BASELINE CHARACTERISTICS:
Arm/Group | Patients Will Undergo Donor/Recipient Bone Marrow
Number analyzed (Participants) | 44
Age, Continuous [Median (Full Range); unit: years] | 62 [35 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 25
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Undergoing an Allo HCT Transplant Who Have a KIR Favorable Donor.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Will Undergo Donor/Recipient Bone Marrow
Number analyzed (Participants) | 44
Participants
  Pts with KIR favorable donor | 23
  Pts without KIR favorable donor | 21

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Patients Will Undergo Donor/Recipient Bone Marrow
All-Cause Mortality (participants affected / at risk) | 17/44
Serious Adverse Events (participants affected / at risk) | 10/44
Other Adverse Events (participants affected / at risk) | 43/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Will Undergo Donor/Recipient Bone Marrow (N=44)
Acute kidney injury (Renal and urinary disorders) | 3
Allergic reaction (Immune system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bronchial infection (Infections and infestations) | 1
Delirium (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Kidney infection (Infections and infestations) | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Lung infection (Infections and infestations) | 4
Myocardial infarction (Cardiac disorders) | 1
Neutrophil count decreased (Investigations) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Sepsis (Infections and infestations) | 5
Small intestine infection (Infections and infestations) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vestibular disorder (Ear and labyrinth disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Will Undergo Donor/Recipient Bone Marrow (N=44)
Abdominal Pain (Gastrointestinal disorders) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Alanine aminotransferase increased (Investigations) | 4
Anemia (Blood and lymphatic system disorders) | 27
Anorexia (Metabolism and nutrition disorders) | 1
Aspartate aminotransferase increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 3
Colitis (Gastrointestinal disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 23
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2
Hyperuricemia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 15
Hypokalemia (Metabolism and nutrition disorders) | 17
Lymphocyte count decreased (Investigations) | 43
Nausea (Gastrointestinal disorders) | 1
Neutrophil count decreased (Investigations) | 28
Pain (General disorders) | 3
Platelet count decreased (Investigations) | 43
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Sepsis (Infections and infestations) | 1
Vertigo (Ear and labyrinth disorders) | 1
White blood cell decreased (Investigations) | 43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/93/NCT02880293/Prot_SAP_000.pdf